CLINICAL TRIAL: NCT05628311
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study (DREAMS-1) to Evaluate the Efficacy and Safety of IBI362 in Chinese Type 2 Diabetes Patients With Poor Glycemia Control Only Through Diet and Exercise
Brief Title: A Study of IBI362 in Poorly Controlled Type 2 Diabetes Patients Only Through Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362A301
Record Dates: First submitted 2022-11-17; First posted 2022-11-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI362 4.0 mg (Experimental): ①2mg, subcutaneously (SC), once a week* 4weeks;
  ②4mg, SC, once a week* 44weeks.
  Interventions: Drug: IBI362
- IBI362 6.0 mg (Experimental): ①2mg, SC, once a week* 4weeks;
  ②4mg, SC, once a week* 4weeks；
  ③6mg, SC, once a week* 40weeks.
  Interventions: Drug: IBI362
- placebo (Placebo Comparator): * placebo, SC, once a week* 24weeks;
    * 2mg, SC, once a week* 4weeks;
      * 4mg, SC, once a week* 4weeks；
        * 6mg, SC, once a week* 16weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — placebo administered subcutaneously (SC) once a week.
  Arms: placebo
Drug: IBI362 — IBI362 administered subcutaneously (SC) once a week.
  Arms: IBI362 4.0 mg; IBI362 6.0 mg

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to evaluate the effectiveness and safety of IBI362 in patients with type 2 diabetes (T2D) with poor glycemia control only through diet and exercise. This study plans to enroll about 300 T2D subjects who still fail to meet the HbA1c standard after at least 2 months of simple diet and exercise control. During the whole study, subjects will be required to maintain diet and exercise control.

The whole trial period includes a 2-week screening period, a 6-week introduction period, a 24 week double-blind treatment period, a 24 week study extension period and a 4-week safety follow-up period.

Subjects who met the randomization criteria will be randomly assigned to the IBI362 4.0 mg group, the IBI362 6.0 mg group and the placebo group at 1:1:1. The randomization stratification factors were (V3) HbA1c<8.5% or HbA1c ≥ 8.5% before randomization.

ELIGIBILITY:
Inclusion Criteria:

1. T2D was diagnosed according to WHO standards in 1999 for at least 2 months
2. Age ≥ 18 when signing the informed consent form
3. The blood glucose was not well controlled after simple diet and exercise within 2 months before screening, and the local laboratory tested 7.5% ≤ HbA1c ≤ 10.5% during screening
4. Maintain a stable diet and exercise lifestyle during the study
5. Subjects voluntarily signed the informed consent form and agreed to strictly follow the requirements of this protocol

Exclusion Criteria:

1. Subjects who the investigator thinks may be allergic to the components in the study drug or similar drugs
2. Weight change>5% within 12 weeks before screening (chief complaint)
3. Used any oral hypoglycemic drugs within 2 months before screening; ≥ 3 oral hypoglycemic drugs have been used together more than 2 months before screening
4. Previous diagnosis of type 1 diabetes (including adult latent autoimmune diabetes), special type diabetes or gestational diabetes
5. There are active or untreated malignant tumors within 5 years before screening, or patients are in remission of clinical malignant tumors (except patients with skin basal cell carcinoma and squamous cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or papillary thyroid carcinoma who have no recurrence after surgery)
6. Mental illness existed in the past or at the time of screening, and the researcher thinks it is not suitable to participate in this study
7. Pregnant or lactating women, or men or women who are fertile and unwilling to use contraception throughout the study period
8. The investigator believes that the subject has any other factors that may affect the efficacy or safety evaluation of this study and is not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline at week 24 | Baseline, 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c<7.0% at week 24 | Baseline, 24 weeks
Safety, Incidence and severity of adverse events and correlation with study drug; | Baseline to 52 weeks
Time to peak plasma concentration (Tmax) | Baseline to 52 weeks
Time to peak plasma concentration (Cmax) | Baseline to 52 weeks
area under curve (AUC) | Baseline to 52 weeks
volume distribution (V) | Baseline to 52 weeks
half-life (half-life, T1/2) | Baseline to 52 weeks
clearance rate (clearance, CL) | Baseline to 52 weeks
To assess changes in PD parameters fasting insulin at different time points before and after administration. | Baseline to 52 weeks
To assess changes in PD parameters fasting C-peptide at different time points before and after administration. | Baseline to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No